CLINICAL TRIAL: NCT02364180
Title: Electromyography With Repetitive Nerve Stimulation in Patients on Chronic Pyridostigmine Therapy
Brief Title: Electromyography in Patients on Chronic Pyridostigmine Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Bhatt Pyriodostigmine
Record Dates: First submitted 2014-12-09; First posted 2015-02-16 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Electromyography

STUDY DESIGN:
Intervention Model Description: All subjects taking Pyridostigmine for at least 6mo, except for myasthenia gravis patients, will be considered for the study.Those that participate will answer a few questions pertaining to their medical history and will then undergo electromyography (CMAP) measurement with repetitive stimulation at 2 sites (ulnar nerve at the wrist and the accessory nerve in the neck). The first and fifth stimuli are delivered 2 seconds apart. Eight percent or greater decrement in the CMAP response on repetitive stimulation will be considered positive.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electromyography (Other): Subjects taking pyridostigmine bromide for more than 6 weeks for a condition other than myasthenia gravis were observed with Electromyography (EMG)
  Interventions: Diagnostic Test: Electromyography (EMG)

INTERVENTIONS:
Diagnostic Test: Electromyography (EMG)

SUMMARY:
We intend to measure evoked EMG at two sites in subjects who are chronically taking pyridostigmine.

DETAILED DESCRIPTION:
The investigators are intending to enroll Patients who are chronically treated with pyridostigmine for the treatment of any medical condition and presenting at the investigators' outpatient clinics for follow up appointment. Subjects taking pyridostigmine for the treatment of myasthenia gravis will be excluded. Both adults and children older than 12 years of age will be approached. Those subjects that agree to participate will be asked to sign an informed consent. For the participation of minors a parental (or guardian) consent and subject assent will be obtained. Those that participate will answer a few questions pertaining to their medical history and will then undergo electromyograph (CMAP) measurement with repetitive stimulation at 2 sites (ulnar nerve at the wrist and the accessory nerve in the neck). Evoked electromyogram will be recorded on a computer hard drive. Eight percent or greater decrement in the CMAP response on repetitive stimulation will be considered positive.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been taking pyridostigmine for the treatment of any condition other than myasthenia gravis

Exclusion Criteria

* Subjects taking pyridostigmine for the treatment of myasthenia gravis will be excluded.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shashi Bhatt, MD, Principal Investigator — The University of Toledo
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects taking Pyridostigmine for at least 6months, except for the treatment of myasthenia gravis, will be considered. Subjects will be recruited from existing patients treated at the university and will be seen in the outpatient clinics.
Groups:
- Pyridostigmine Bromide Treatment Group: pyridostigmine bromide treatment is a single arm. Subjects must be treated with pyridostigmine for at least 6months and must not be treated for myasthenia gravis.
Period: Overall Study
Arm/Group | Pyridostigmine Bromide Treatment Group
Started | 11
Completed | 10
Not Completed | 1
Not completed — Screen Fail | 1

BASELINE CHARACTERISTICS:
Groups:
- Pyridostigmine Bromide Treatment Group: All subjects investigated were taking pyridostigmine.
Arm/Group | Pyridostigmine Bromide Treatment Group
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 63 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Amplitude of Evoked Compound Muscle Action Potential by Electromyography Between the First to Fifth Response
Description: Normally when a nerve is rapidly stimulated the successive Compound Muscle Action Potentials (CMAP) are of the same height. We are hoping to investigate if chronic pyridostigmine therapy reduces the margin of safety and hence the successive CMAPs may be smaller than the preceding ones.
Time Frame: Baseline measurement only. First and Fifth stimuli delivered 2 seconds apart on the same day. There are no additional days/times.
Measure: Median (Full Range); unit: percent change
Groups:
- Pyridostigmine Bromide Treatment Group: Subjects taking pyridostigmine bromide for more than 6 months for a condition other than myasthenia gravis
Arm/Group | Pyridostigmine Bromide Treatment Group
Number analyzed (Participants) | 10
percent change | 0 [-4 to 13]

ADVERSE EVENTS:
Time Frame: There were no adverse events to collect during the time of the subject participation which was 1 day.
Groups:
- Pyridostigmine Bromide Treatment Group: In all enrolled subjects (10), who were known pyridostigmine bromide pts that were observed with Electromyography (EMG), there were no adverse events anticipated.
Arm/Group | Pyridostigmine Bromide Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes